CLINICAL TRIAL: NCT01006447
Title: Tai Chi/Qigong Exercise Persistence Among Residents of Senior Housing: a Randomized Field Trial
Brief Title: Tai Chi/Qigong Exercise Persistence Among Residents of Senior Housing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: D'Youville College (Other)
Collaborators: Community Health Foundation Western NY (Unknown); People. Inc (Unknown)
Responsible Party: Peneolpe J. Klein, D'Youville College
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DYC-023
Record Dates: First submitted 2009-11-01; First posted 2009-11-02 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-11

CONDITIONS: Physical Activity
Keywords: tai chi; exercise; older adults; exercise persistence
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Instructor contact 1 class (Active Comparator)
  Interventions: Behavioral: Instructor contact
- Instructor contact 4 classes (Active Comparator)
  Interventions: Behavioral: Instructor contact

INTERVENTIONS:
Behavioral: Instructor contact
  Arms: Instructor contact 1 class
Behavioral: Instructor contact
  Arms: Instructor contact 4 classes

SUMMARY:
This randomized field trial uses a self-report daily exercise log to answer the research question: Does frequency of instruction influence tai chi/qigong home practice exercise persistence among residents of Senior housing?

ELIGIBILITY:
Inclusion Criteria:

* Resident of Senior housing,
* Ability to engage in mild exercise
* Vision sufficient to view TV medium
* Willingness to engage in tai chi/qigong training and practice.

Exclusion Criteria:

* Unable to provide informed consent
* Unable to attend initial training session

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
exercise persistence | 3 months

SECONDARY OUTCOMES:
perceived benefits | 3 months
barriers to exercise | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - D'Youville College, Buffalo, New York
  - People, Inc Senior Housing Buildings, Williamsville, New York